CLINICAL TRIAL: NCT04871984
Title: Ureteroscopy for Upper Tract Lithiasis : Comparison of Costs and Effectiveness of Both Holmium and Thulium Lasers, in a Prospective Monocentric Study.
Brief Title: Effectiveness of Holmium and Thulium Lasers With Ureteroscopy for Urinary Lithiasis
Acronym: LiThuHol
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: ar21-0020v0
Record Dates: First submitted 2021-02-25; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Renal Stone; Ureteral Stone
MeSH Terms: conditions — Nephrolithiasis; Ureterolithiasis | interventions — Ureteroscopy; Lasers, Solid-State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Holmium laser lithotripsy: Stone fragmentation are performed with Holmium laser in ureteroscopy
  Interventions: Device: Ureteroscopy for upper tract stone treatment with Holmium laser
- Thulium laser lithotripsy: Stone fragmentation are performed with Thulium laser in ureteroscopy
  Interventions: Device: Ureteroscopy for upper tract stone treatment with Thulium laser

INTERVENTIONS:
Device: Ureteroscopy for upper tract stone treatment with Holmium laser — Rigid or flexible ureteroscopy for ureteral or renal stone. Lithotripsy with Holmium laser
  Groups: Holmium laser lithotripsy
Device: Ureteroscopy for upper tract stone treatment with Thulium laser — Rigid or flexible ureteroscopy for ureteral or renal stone. Lithotripsy with Thulium laser
  Groups: Thulium laser lithotripsy

SUMMARY:
Holmium laser is the current gold standard for lithotripsy on urinary lithiasis, while Thulium is brand new. The latter has been released in July 2020 in Europe, and only in-vitro studies have been published.

The aim of this study is to compare the stone free rate in ureteroscopy, for all consecutive patients treated with laser fragmentation, between both Holmium and Thulium lasers.

The costs and complications will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* renal ou ureteral stone confirmed by an abdominal and pelvic computed tomography
* treatment with rigid or flexible ureteroscopy
* laser lithotripsy during the procedure
* bacteriological examination of urine (sterile, bacterial colonization or treated by antibiotics)

Exclusion Criteria:

* non-use of laser for stone lithotripsy
* pregnant women
* under 18 years old
* refusal to give informed consent
* urinary malformation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled for ureteroscopy on renal or ureteral stones, which have been previously confirmed by tomography
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Stone free rate | Three months after surgery
  Urinary tract echography or renal computer tomography imaging. Patients with residual fragments under 4 mm are stone free.

SECONDARY OUTCOMES:
Perioperative complications | During the intervention
  Recording data about ureteric perforation and bleeding
Operating time | Immediately after the intervention
  All surgeries are included
Postoperative complications | Up to three months after surgery
  Recording data according to the Clavien classification (rates of hospitalisation, pain, infection and surgical revision)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Panthier F, Doizi S, Corrales M, Traxer O. Pulsed lasers and endocorporeal laser lithotripsy. Prog Urol. 2021 Jun-Jul;31(8-9):451-457. doi: 10.1016/j.purol.2020.11.008. Epub 2021 Jan 28. PMID 33516610
- [Background] Martov AG, Ergakov DV, Guseinov MA, Andronov AS, Dutov SV, Vinnichenko VA, Kovalenko AA. [Initial experience in clinical application of thulium laser contact lithotripsy for transurethral treatment of urolithiasis]. Urologiia. 2018 Mar;(1):112-120. Russian. PMID 29634144
- [Background] Rapoport LM, Vinarov AZ, Sorokin NI, Dymov AM, Enikeev DV, Tsarichenko DG, Lekarev VY, Klimov RE, Andreeva VA, Kovalenko AA. [Experimental verification of thulium lithotripsy]. Urologiia. 2018 Dec;(5):74-80. Russian. PMID 30575354